CLINICAL TRIAL: NCT05805046
Title: Postmarket Clinical Follow-Up Study of Avelle™ Negative Pressure Wound Therapy (NPWT) System in Patients With Acute Wounds
Brief Title: Study of Avelle™ Negative Pressure Wound Therapy (NPWT) System
Status: Withdrawn | Type: Observational
Why Stopped: Convatec has identified an external source that has already collected relevant real-world data in a manner consistent with the proposed clinical study objectives.
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: WC22431
Record Dates: First submitted 2023-03-28; First posted 2023-04-07 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Surgical Wound, Recent; Surgical Wound Leak; Dehiscence Wound; Trauma-related Wound
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Negative Pressure Wound Therapy System — The study device combines a sterile dressing comprising gelling fibre technology to absorb wound exudate with negative pressure applied to the wound via a vacuum pump.
  Other Names: Avelle™ Negative Pressure Wound Therapy System

SUMMARY:
The main questions the study aims to answer are:

* How much do wounds improve when using the Avelle™ Negative Pressure Wound Therapy System for a maximum of 14 days?
* How safe is the Avelle™ Negative Pressure Wound Therapy System?

DETAILED DESCRIPTION:
The goal of this observational study is to gather information about the the Avelle™ Negative Pressure Wound Therapy System in people that have a wound that leaks fluid and is 14 days old or less. The Avelle™ Negative Pressure Wound Therapy (NPWT) System combines a sterile dressing comprising gelling fibre technology to absorb wound exudate with negative pressure applied to the wound via a vacuum pump. The Avelle™ NPWT System consists of a disposable single patient use battery powered pump, absorbent wound dressing, and fixation strips.

Participants will:

* be asked questions about their medical history and medications
* asked to allow the wound and surrounding skin to be examined
* be asked to use the Avelle™ Negative Pressure Wound Therapy System for a maximum of 14 days
* be asked to review any issues or concerns with the Avelle™ Negative Pressure Wound Therapy System

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age.
2. Subject is willing and able to take part in the study and provide written informed consent.
3. Subject has one target wound which is ≤ 14 days old
4. Subject has target wound that is intended to heal by primary intention
5. Subject has a target wound which is ≤ 25% of the dressing area as per the Instructions For Use
6. Target wound has low to moderate exudate
7. Wound is suitable for treatment with Avelle™ NPWT
8. Subject is deemed capable and willing to comply with the protocol and product instructions.

Exclusion Criteria:

1. Subject has an existing health condition that would compromise their participation and follow-up in this study such as the ability to understand and follow instructions
2. Subject has been treated with another NPWT system during the past 14 days
3. Subject, in the opinion of the Investigator, is not clinically suitable for inclusion
4. Subject is contraindicated for the Avelle™ NPWT System

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Negative pressure wound therapy is used to assist in the management of a closed surgical wound or other acute wound expected to heal by way of primary intention.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Complete wound healing evidenced by substantially complete epithelialization (>95% by area estimate). | Up to 14 days
  Primary performance outcome
Frequency of device-related serious adverse events (SAEs) (all adverse events attributed to the wound and or device will be collected and assessed as non-device related or device related, and serious or non-serious, by the Investigator) | Up to 14 days
  Primary safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Cristin Taylor, Study Director — AWC Senior Director, Convatec
Locations (4):
- United States (4):
  - The Angel Medical Research Corp, Miami Lakes, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Northwell Health, Lake Success, New York
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No